CLINICAL TRIAL: NCT02882009
Title: A Single-Center, Randomized, Open-Label, Parallel-Group, Placebo-Controlled, Cross-Over Study To Investigate the Impact of Speed of Injection and Site of Injection on Pain, Tolerability, Safety, and Pharmacokinetics Following Subcutaneous Administration of Gantenerumab in Healthy Volunteers
Brief Title: A Study to Assess the Impact of Speed and Site of Subcutaneous Injection on Pain, Tolerability, Safety, and Pharmacokinetics of Gantenerumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP39322
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gantenerumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gantenerumab + Placebo (Experimental): Participants will be randomized to receive gantenerumab HCLF and placebo solution via SC injection according to different sequences for the site of administration and different injection speeds.
  Interventions: Drug: Gantenerumab; Drug: Placebo

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab as a HCLF will be administered via SC injection according to assigned treatment sequence.
  Other Names: RO4909832
Drug: Placebo — Gantenerumab Placebo solution will be administered via SC injection according to assigned treatment sequence.

SUMMARY:
The purpose of this randomized, open-label, parallel-group, placebo-controlled study is to assess pain following subcutaneous (SC) administration of gantenerumab as a high-concentration liquid formulation (HCLF) at different injection speeds. The total duration of the study for each healthy participant will be up to approximately 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants (healthy status is defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram, hematology, blood chemistry, coagulation, serology, and urinalysis)
* Body mass index between 18.0 and 30.0 kilograms per meter squared (kg/m^2), inclusive
* Female participants of childbearing potential must commit to use two acceptable forms of contraception during the study and until at least 6 months after the follow-up visit

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer, or cirrhosis
* History or suspicion of drugs of abuse or alcohol addiction
* Smokers who smoke more than 10 cigarettes per day or equivalent amount of tobacco as determined by history
* Pregnant or lactating women
* Positive result on hepatitis B virus (HBV), hepatitis C virus (HCV), or Human immunodeficiency virus (HIV)-1 and -2
* Any familial history of early onset Alzheimer's disease
* Prior administration of gantenerumab
* Participation in an investigational drug medicinal product or medical device study within 90 days before dosing or within seven times the elimination half-life, whichever is longer
* Any abnormal skin conditions or potentially obscuring tattoos, pigmentation, or lesions in the area intended for SC injection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-08-31 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Local Pain as Assessed Using Visual Analog Scale (VAS) | Immediately after the injection on Day 1

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Gantenerumab | 0 hour (predose) and 6, 12, and 24 hours postdose on Day 1, on Days 2, 3, 4, 5, 6, 7, 8, 12, 21, 43, 64, 85
Area Under the VAS Pain-Time Curve From Time 0 to 20 Minutes (AUC[0-20]) | 0 to 20 minutes after injection on Day 1
Local Pain as Assessed Using Verbal Rating Scale (VRS) Score | Immediately after the injection on Day 1
Number of Participants With Skin Reactivity, as Assessed Using a 0 (No Reactivity) to 3 (Severe Reactivity) Scale | Immediately post-dose to 6 hours on Day 1
Number of Participants With Adverse Events | From Screening to Day 85
Number of Participants With Anti-Gantenerumab Antibodies (ADAs) | Day 1 (predose [Hour 0]) and Day 85
Maximum Observed Plasma Concentration (Cmax) of Gantenerumab | 0 hour (predose) and 6, 12, and 24 hours postdose on Day 1, on Days 2, 3, 4, 5, 6, 7, 8, 12, 21, 43, 64, 85

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA International Clinical Pharmacology Center (EDS US Clinic), Lenexa, Kansas, United States

REFERENCES:
- [Derived] Portron A, Jordan P, Draper K, Muenzer C, Dickerson D, van Iersel T, Hofmann C. A Phase I Study to Assess the Effect of Speed of Injection on Pain, Tolerability, and Pharmacokinetics After High-volume Subcutaneous Administration of Gantenerumab in Healthy Volunteers. Clin Ther. 2020 Jan;42(1):108-120.e1. doi: 10.1016/j.clinthera.2019.11.015. Epub 2019 Dec 26. PMID 31883703